CLINICAL TRIAL: NCT05899088
Title: A Randomized Clinical Trial of Mindful Movement for Patients With Chronic Pelvic
Brief Title: Mindful Movement for Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: Rhode Island Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1979873; 7141745 (Other Grant/Funding Number: Rhode Island Foundation)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Pelvic Pain; Endometriosis
Keywords: Chronic Pelvic Pain, Kinesiophobia, Mindful movement, Endometriosis
MeSH Terms: conditions — Pelvic Pain; Endometriosis; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Rolling admission of participants. Each participant completes 12 weeks of intervention with weekly follow-up if in treatment arm. No follow-up in control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Patients follow-up as normal with physician. Recommended by physician to engage in physical activity 4x/w. No other intervention or follow-up.
- Study Arm (Experimental): Patients engage in weekly exercise program as recommended by the study. Researchers follow up weekly with patient to assess progress. Complete surveys at beginning and end.
  Interventions: Other: Mindful Movement

INTERVENTIONS:
Other: Mindful Movement — Mindful Movement Program with Researcher Follow-up
  Arms: Study Arm

SUMMARY:
Female chronic pelvic pain (CPP) is defined as the sensation of pain arising from the lower urinary tract, bowel, muscles, nerves, and gynecologic organs within the pelvis. It can also include menstrual pain and pain with intercourse, when these adversely affects a patient's well-being. Chronic pelvic pain is often associated with negative cognitive, behavioral, sexual and emotional consequences, which can include physical deconditioning, pain catastrophizing (magnifying the threat of pain), kinesiophobia (fear of movement), and depression. CPP has been estimated to affect between 5.7%-26.6% of women.Treatments for chronic pelvic pain are limited, and the use of centrally acting pain medications such as opioids is common. There is increasing awareness of the risks of these medications, including dependence, addiction, and over-dose related death. Therefore, it is critical to look for safe alternatives to manage chronic pelvic pain.

Exercise has been targeted as a treatment strategy for chronic pain conditions, improving both pain intensity and physical function. Studies have demonstrated that yoga, Zumba®, and treadmill walking can improve menstrual related pain and quality of life. Mindfulness is the non-judgmental acceptance and investigation of present experience, including body sensations, internal mental states, thoughts, emotions, impulses, and memories to reduce suffering or distress and to increase well-being. Prior research by our group has demonstrated efficacy of mindfulness meditation in reducing pain and improving quality of life in women with chronic pelvic pain. Mindful movement is putting attention into what the body is feeling as it moves. It involves paying attention movement that feels good as well as to early warning signs that an exercise may be too intense or may cause a pain flare.

This study is a 12-week program of gentle aerobic exercise and stretching for patients with CPP that applies mindful movement practices. Patients will be randomized to weekly classes versus the routine recommendations for exercise. We will measure pain reduction, improvement in quality of life, and reduction in pain catastrophizing and kinesiophobia.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is defined as the sensation of pain arising from the lower urinary tract, bowel, pelvic floor, myofascial, and reproductive structures and includes cyclic pain and pain with intercourse, when the condition adversely affects a patient's wellbeing. Chronic pelvic pain is often associated with negative cognitive, behavioral,sexual and emotional consequences, which can include physical deconditioning, pain catastrophizing, kinesiophobia, and depression. CPP has been estimated to affect between 5.7%-26.6% of women.

Treatments for pelvic pain include management of peripheral pain sources, as well as targeting the centrally mediated response to pain. The use of centrally acting pain medications, including opioids, is common in patients with pelvic pain. There is increasing literature recommending against the use of opioids for chronic pain, citing risks of dependence, addiction, and over-dose related death. Therefore, it is critical to look for safe alternatives to manage chronic pelvic pain.

Exercise has been targeted as a treatment strategy for chronic pain conditions, improving both pain intensity and physical function. Multiple studies have demonstrated that yoga, Zumba®, and treadmill walking can improve menstrual-related pain in young women with dysmenorrhea. In addition to pain reduction, studies have also demonstrated improvement in quality of life. Mindfulness is the non-judgmental acceptance and investigation of present experience, including body sensations, internal mental states, thoughts, emotions, impulses, and memories to reduce suffering or distress and to increase well-being. Prior research by our group has demonstrated efficacy of mindfulness meditation in reducing pain and improving quality of life in women with chronic pelvic pain. Mindful movement is putting attention into what the body is feeling as it moves. It involves paying attention movement that feels good as well as to early warning signs that an exercise may be too intense or may cause a pain flare.

This study is a 12-week program of aerobic exercise and stretching for patients with CPP that applies mindful movement practices. Patients will be randomized to weekly classes versus routine recommendations for exercise. We will measure pain reduction, improvement in quality of life, and reduction in pain catastrophizing and kinesiophobia.

We will enroll patients with chronic pelvic pain of at least 6-months duration who have not engaged in regular physical activity in the prior 3 months. Patients aged 18 or older receiving care in the Pelvic Pain Program at the WMC will be invited to take part in the study. Records for patients in the pelvic pain program who are presenting for care will be reviewed for eligibility and approached prior to their visit about potentially participating in the study. Additionally, charts for patients active in the pelvic pain program will be reviewed for eligibility and the research assistant contact participants about participation in the study. If patients are interested in the study and do not have an upcoming office visit, they will be scheduled to come in to meet with the research assistant and be consented for the study. Subjects will also be consented at the time of their office visits.

Study methods:

1. 60 patients with a history of CPP who meet the inclusion and exclusion criteria will be recruited and randomly assigned to the mindful movement program (N=30) or routine care (N=30).
2. All subjects will watch a video, created by our program for the pelvic pain population, which will review safety measures for starting an exercise program. The video includes how to start and gently increase duration of exercise and modifications that can be used to safely exercise with pain. All subjects will receive a step tracker and a study journal.
3. Patients randomized to the study arm will get a prescription for aerobic mindful exercise and stretching 4 days a week. They will view additional videos, created by our program, about mindful movement, awareness of body cues, intentional movement, and body scans. The scripts for the videos are submitted to the IRB for approval. They will have access to exercise classes as described below that are geared toward participants with physical limitations. All classes will incorporate reminders regarding mindful movement practices, as teachers will be selected who have an understanding of this principle. Participants will be instructed to attend an in person or virtual class at least once a week. A variety of 20-60 minute classes will be available. Participants will be reminded to listen to their body's cues and be given options to modify their movement. Additionally, participants will work towards completing at least 20 minutes of walking followed by 5-10 minutes of stretching 3 days a week. Participants can attend additional classes instead of walking. Participants are instructed to work toward a goal of at least. 80 minutes of cardiovascular exercise along with stretching each week. Participants will be required to track their activity with a study journal and step tracker provided through the study.

   a. Walking exercise with stretching: Participants will be recommended to walk on a treadmill, outside, or indoor location for at least 20 minutes, at a pace brisk enough to elevate ones heart rate. Participants are instructed to gently stretch their muscles following this activity for approximately 5-10 minutes.

   b. Yoga is a physical and mental practice with ancient roots. Modern yoga generally intends to build strength, stamina, flexibility, coordination and balance through a series of poses.

   c. Shake your Soul® is a movement practice that was developed with mindfulness practices in mind. It incorporates fluid dance repertoire set to world music. Classes cannot be recorded.

   d. Zumba® is a dance exercise class that features Latin and World rhythms. It provides a total workout, combining cardio, muscle conditioning, balance, and flexibility. Lower impact versons, such as Zumba Gold® have been designed to meet the needs of seniors and others who need lower impact activity. Classes cannot be recorded
4. Weekly phone calls with the research assistant will include collection of pain scores and will review barriers to exercise, pain issues related to the exercise and mindful approach to exercise. If a participant feels they may have an injury or are unable to continue the program, Dr. Clark Donat or Dr. Fox will be notified and follow up accordingly.
5. Patients randomized to the control arm will receive routine care within the pelvic pain program. As part of routine care, patients are counseled on the importance of movement and encouraged to engage in gentle activity. They will be given access to the introductory video. Participants will be encouraged to walk or engage in some form of cardiovascular exercise for at least 20 minutes a day, 4 days a week, and gently stretch for 5-10 minutes after their exercise. Participants are instructed to increase work toward a goal of at least. 80 minutes of cardiovascular exercise along with stretching each week. Participants will be encouraged to reach out to the study team if they feels they may have an injury or are unable to continue the program, Dr. Clark Donat or Dr. Fox will be notified and follow up accordingly.
6. Pain scores will be obtained using an 11-point NPS by the research assistant at the initial visit and during weekly phone check-ins.
7. Quality of life will be assessed using the World Health Organization Quality of Life -BREF questionnaire, a 26-item validated tool that addresses 4 domains: physical health, psychological health, social relationships, and environmental health [21]. Kinesiophobia will be assessed using the validated Tampa Scale for Kinesiophobia, a 17-item tool that indicates the level of fear associated with movement [22]. Pain catastrophizing will be assessed using the Pain Catastrophizing Scale, a validated 13- item tool that examines three subscales: magnification, rumination and helplessness [23]. These tools will be administered at enrollment and week 12.
8. Patient charts will be reviewed for demographics information, pain diagnoses and treatments, and medical and surgical history.

Summary Study Outline following randomization

Study Arm (1) vs. Control Arm (2) Initial exercise video

1. Yes- prior to initiation of 12 week program 2. Yes- prior to initiation of 12 week program Step tracker and study journal

1. Yes- prior to initiation of 12 week program
2. Yes- prior to initiation of 12 week program Mindful Movement video

1. Yes- prior to initiation of 12 week program 2. No Prescription for weekly exercise

1. Yes- 4 days a week with a goal of 80 minutes of cardiovascular exercise plus stretching a week: including at least one class
2. No, but participants will be encouraged to exercise 4 days a week with a goal of 80 minutes of cardiovascular exercise plus stretching each week.

Weekly Phone calls by research assistant

1. Yes- with follow up by Drs. Clark Donat or Fox as indicated
2. No Assessment of Pain scores

1. Yes- at intake and weekly by RA 2. Yes- at intake and at conclusion of study Questionnaires

1. Yes- At enrollment and week 12 via RedCap
2. Yes- At enrollment and week 12 via RedCap

Benefits:

Study subjects may benefit from improved pain levels, improved quality of life, and increased fitness level. They may also benefit from developing increased insight about how movement helps their pain and how to understand their bodies signal in relationship to exercise.

Risks:

There is limited risk to the subjects who choose to participate in this study. All recruited patients will already be undergoing care for their chronic pelvic pain, and therefore being counseled generally on the importance of gentle exercise and movement. New exercise can be associated with musculoskeletal soreness or injury, some participants may notice changes in their bowel or bladder habits, and participants could experience dehydration. To minimize these risks and prepare participants for these side effects, the exercise will be slow and gentle with incorporated stretching, participants will be counseled on adequate hydration, and made aware that bowel and bladder changes may be encountered. As part of the weekly check in calls the research assistant will screen for possible side effects from exercise and provide appropriate information or alter the providers to contact the patient.

Potential Obstacles:

Studies of patients with CPP often have a low completion rate because of chronic pain and life stressors [16]. We hope that this program of mindful movement, with a slow and gentle increase in duration, will help to allow more subjects to continue this program. In addition, we will be providing a small stipend to help encourage completion of the study. Since much of the exercise will be available virtually, there may be a barrier with poor access to the internet. However, patients will be given the option of a walking program that can be completed independently. Lastly, pain catastrophizing and kinesiophobia may also be barriers for this study. We hope that our gentle approach to exercise will allow patient to engage in the program. Additionally, we will monitor patient experience with pain catastrophizing and kinesiophobia as a study outcome.

Confidentiality of Data:

Medical records of all patients enrolling in the study will be reviewed for demographic and health related information. Protected Health Information (PHI) obtained will include patient's name and date of birth. Additionally, information from the questionnaires will be obtained. All information will be kept in a REDCAP database. Responses to the questionnaires will be put into the database, and all hard copies will be discarded. After data collection is complete, all data will be de-identified and a key to allow the information to be linked to the appropriate patient will be kept in a separate, password-protected database on a Lifespan computer. The de-identified database will be used for statistical analysis and presentation of data to the team, in order to maintain HIPPA compliance. Hard copies of the consent forms will be kept in a locked file cabinet in Dr. Sarah Fox's office. The final data will be analyzed and published in a group format, and will not be traceable to specific patients. No information about sensitive or illegal behavior will be obtained.

Participate compensation:

All subjects will be given a fitness tracker valued at $30, They will also be compensated $25 for completion of the surveys at 6 and 12 weeks. Additionally, participants who are randomized to the study arm will receive access to virtual and in person exercise classes free of charge.

Timeline:

In preparation for this application, the PI reviewed records of the patients seen in the Pelvic Pain Program for the month of September 2021. 27 patients seen in that month would have been eligible for the study. For this reason, we are confident that we would be able to recruit and randomize our target of 60 patients within 6 months of beginning recruitment. Research Team:The investigators all have extensive experience caring for patients with chronic pain conditions. We have worked together clinically for up to 12 years and have been actively involved in research on mindfulness for the past 4 years. The current research team previously studied mindfulness meditation for CPP so they have experience with this patient population and have already established successful collaboration [16].

ELIGIBILITY:
Inclusion Criteria:

* Must receive care in the Pelvic Pain Program at the Women's Medicine Collaborative at Lifespan
* Aged 18 or over
* Able to ambulate independently
* Not exercising regularly: defined by less than 30 minutes of aerobic exercise per week in the past 3 months.
* Able to speak and understand conversational English. Written materials will be available in English and Spanish.

Exclusion Criteria:

* Under age 18
* Currently pregnant or up to 6 weeks postpartum
* Medical conditions for which exercise is contraindicated
* Major surgery within the past 12 weeks or planned within the next 12 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in Pelvic Pain Level | 12 weeks
  To determine if mindful movement can reduce pain in a patient with CPP
Impact on Quality of Life | 12 weeks
  To determine if mindful movement can improve quality of life in patients with CPP
Change in Kinesiophobia and Pain Catastrophizing | 12 weeks
  To determine if mindful movement can reduce kinesiophobia and pain catastrophizing in patients with CPP

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chronic Pelvic Pain: ACOG Practice Bulletin, Number 218. Obstet Gynecol. 2020 Mar;135(3):e98-e109. doi: 10.1097/AOG.0000000000003716. PMID 32080051
- [Background] American College of Obstetricians and Gynecologists. Revitalize. Gyencology data definitions (version 1.0). Washington, DC: American College of Obstetricians and Gynecologists: 2018. Available at : Httph://www.acog.org/-/media/Departments/patient-safety-and-quality-improvement/revit alize-Gynecology-Definitions-V2.pdf. Retrieved 5/2/2021
- [Background] Ahangari A. Prevalence of chronic pelvic pain among women: an updated review. Pain Physician. 2014 Mar-Apr;17(2):E141-7. PMID 24658485
- [Background] Simoens S, Dunselman G, Dirksen C, Hummelshoj L, Bokor A, Brandes I, Brodszky V, Canis M, Colombo GL, DeLeire T, Falcone T, Graham B, Halis G, Horne A, Kanj O, Kjer JJ, Kristensen J, Lebovic D, Mueller M, Vigano P, Wullschleger M, D'Hooghe T. The burden of endometriosis: costs and quality of life of women with endometriosis and treated in referral centres. Hum Reprod. 2012 May;27(5):1292-9. doi: 10.1093/humrep/des073. Epub 2012 Mar 14. PMID 22422778
- [Background] Steege JF, Siedhoff MT. Chronic pelvic pain. Obstet Gynecol. 2014 Sep;124(3):616-629. doi: 10.1097/AOG.0000000000000417. PMID 25162265
- [Background] As-Sanie S, Soliman AM, Evans K, Erpelding N, Lanier RK, Katz NP. Short-acting and Long-acting Opioids Utilization among Women Diagnosed with Endometriosis in the United States: A Population-based Claims Study. J Minim Invasive Gynecol. 2021 Feb;28(2):297-306.e2. doi: 10.1016/j.jmig.2020.05.029. Epub 2020 Jun 9. PMID 32531340
- [Background] Rosenberg JM, Bilka BM, Wilson SM, Spevak C. Opioid Therapy for Chronic Pain: Overview of the 2017 US Department of Veterans Affairs and US Department of Defense Clinical Practice Guideline. Pain Med. 2018 May 1;19(5):928-941. doi: 10.1093/pm/pnx203. PMID 29025128
- [Background] Geneen LJ, Moore RA, Clarke C, Martin D, Colvin LA, Smith BH. Physical activity and exercise for chronic pain in adults: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2017 Apr 24;4(4):CD011279. doi: 10.1002/14651858.CD011279.pub3. PMID 28436583
- [Background] Rakhshaee Z. Effect of three yoga poses (cobra, cat and fish poses) in women with primary dysmenorrhea: a randomized clinical trial. J Pediatr Adolesc Gynecol. 2011 Aug;24(4):192-6. doi: 10.1016/j.jpag.2011.01.059. Epub 2011 Apr 21. PMID 21514190
- [Background] Yang NY, Kim SD. Effects of a Yoga Program on Menstrual Cramps and Menstrual Distress in Undergraduate Students with Primary Dysmenorrhea: A Single-Blind, Randomized Controlled Trial. J Altern Complement Med. 2016 Sep;22(9):732-8. doi: 10.1089/acm.2016.0058. Epub 2016 Jun 17. PMID 27315239
- [Background] Yonglitthipagon P, Muansiangsai S, Wongkhumngern W, Donpunha W, Chanavirut R, Siritaratiwat W, Mato L, Eungpinichpong W, Janyacharoen T. Effect of yoga on the menstrual pain, physical fitness, and quality of life of young women with primary dysmenorrhea. J Bodyw Mov Ther. 2017 Oct;21(4):840-846. doi: 10.1016/j.jbmt.2017.01.014. Epub 2017 Feb 7. PMID 29037637
- [Background] Heidarimoghadam R, Abdolmaleki E, Kazemi F, Masoumi SZ, Khodakarami B, Mohammadi Y. The Effect of Exercise Plan Based on FITT Protocol on Primary Dysmenorrhea in Medical Students: A Clinical Trial Study. J Res Health Sci. 2019 Aug 24;19(3):e00456. PMID 31586377
- [Background] Kannan P, Chapple CM, Miller D, Claydon-Mueller L, Baxter GD. Effectiveness of a treadmill-based aerobic exercise intervention on pain, daily functioning, and quality of life in women with primary dysmenorrhea: A randomized controlled trial. Contemp Clin Trials. 2019 Jun;81:80-86. doi: 10.1016/j.cct.2019.05.004. Epub 2019 May 7. PMID 31071464
- [Background] Samy A, Zaki SS, Metwally AA, Mahmoud DSE, Elzahaby IM, Amin AH, Eissa AI, Abbas AM, Hussein AH, Talaat B, Ali AS. The Effect of Zumba Exercise on Reducing Menstrual Pain in Young Women with Primary Dysmenorrhea: A Randomized Controlled Trial. J Pediatr Adolesc Gynecol. 2019 Oct;32(5):541-545. doi: 10.1016/j.jpag.2019.06.001. Epub 2019 Jun 11. PMID 31195099
- [Background] Luque-Suarez A, Martinez-Calderon J, Falla D. Role of kinesiophobia on pain, disability and quality of life in people suffering from chronic musculoskeletal pain: a systematic review. Br J Sports Med. 2019 May;53(9):554-559. doi: 10.1136/bjsports-2017-098673. Epub 2018 Apr 17. PMID 29666064
- [Background] Clark Donat L, Reynolds J, Friedman L, Bublitz M, Flynn E, Fox SD. (2020) October. The Effect of a Brief Mindfulness Meditation Based Intervention on Women with Chronic Pelvic Pain. Poster presentation. 23rdAnnual Scientific Meeting on Pelvic Pain; Virtual.
- [Background] Kabat-Zinn J (2013). Full Catastrophe Living: Using the Wisdom of Your Body and Mind to Face Stress, Pain, and Illness. New York: Bantam Dell. ISBN 978-0345539724.
- [Background] Crane-Okada R, Kiger H, Anderson NL, Carroll-Johnson RM, Sugerman F, Shapiro SL, Wyman-McGinty W. Participant perceptions of a mindful movement program for older women with breast cancer: focus group results. Cancer Nurs. 2012 May-Jun;35(3):E1-10. doi: 10.1097/NCC.0b013e31822539c5. PMID 21897212
- [Background] Chan RR, Larson JL. Meditation Interventions for Chronic Disease Populations: A Systematic Review. J Holist Nurs. 2015 Dec;33(4):351-65. doi: 10.1177/0898010115570363. Epub 2015 Mar 2. PMID 25731777
- [Background] Fox SD, Flynn E, Allen RH. Mindfulness meditation for women with chronic pelvic pain: a pilot study. J Reprod Med. 2011 Mar-Apr;56(3-4):158-62. PMID 21542535
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Miller R, Kori S, Todd D. The Tampa Scale, The Clinical Journal of Pain: March 1991; 7(1):51
- [Background] Sullivan, M. J. L., Bishop, S. R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and validation. Psychological Assessment 1995;7(4):524-32.
- [Background] Safikhani S, Gries KS, Trudeau JJ, Reasner D, Rudell K, Coons SJ, Bush EN, Hanlon J, Abraham L, Vernon M. Response scale selection in adult pain measures: results from a literature review. J Patient Rep Outcomes. 2018 Sep 6;2:40. doi: 10.1186/s41687-018-0053-6. eCollection 2017. PMID 30238085